CLINICAL TRIAL: NCT01200862
Title: An Open-label Dose Finding Study Followed by a Parallel Group, Randomized, Double-blind Study to Evaluate the Safety, Tolerability and Pharmacodynamics of 12 Week BGS649 Treatment in Obese, Hypogonadotropic Hypogonadal Men
Brief Title: Safety and Efficacy of BGS649 in Obese, Hypogonadotropic Hypogonadal Men
Acronym: OHH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Mereo BioPharma (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBGS649A2204
Record Dates: First submitted 2010-09-10; First posted 2010-09-14 (Estimated); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Obese Hypogonadotropic Hypogonadism
Keywords: Obese; obesity; hypogonadism; hypogonadotropic; hyperestrogenemic; testosterone; hypogonadal
MeSH Terms: conditions — Obesity; Hypogonadism

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Open-label in Part 1 and double-blind in Part 2.

ARMS (3):
- BGS649 (Part 1) (Experimental): BGS649 1mg and 0.1mg in hard gelatin capsules. In part 1 there was individualised dosing to titrate the subject's testosterone into the normal range. If the dose was lower than 0.1mg then specific instructions for dilution of an oral solution of BGS649 were provided.
  Interventions: Drug: Investigational new drug company code: BGS649
- Placebo to BGS649 (Part 2) (Placebo Comparator): Matching placebo to BGS649 (0.3 and 0.1mg). 0.3mg placebo capsule given on Day 1 and 0.1mg placebo capsule on other treatment visits (week 1 to 11).
  Interventions: Drug: Placebo
- BGS649 (Part 2) (Experimental): 0.3 or 0.1mg hard gelatin capsules of BGS649 given orally. 0.3mg on Day 1 and 0.1 on all other treatment visits (week 1 to 11).
  Interventions: Drug: Investigational new drug company code: BGS649

INTERVENTIONS:
Drug: Investigational new drug company code: BGS649
  Arms: BGS649 (Part 1); BGS649 (Part 2)
Drug: Placebo
  Arms: Placebo to BGS649 (Part 2)

SUMMARY:
This study is designed as a 2-part study, with Part 1 being open-label to best determine the appropriate dose levels to use in Part 2, which has a randomized, double-blind, placebo controlled design. The study aims to assess the safety and tolerability of BGS649, and determine whether or not BGS649 is able to normalize testosterone levels and improve insulin sensitivity in obese, hypogonadotropic hypogonadal (OHH) men

ELIGIBILITY:
Inclusion Criteria:

* Males who meet the criteria of obese, hypogonadotropic hypogonadism defined as:

  * Patients with a Body Mass Index (BMI) ≥ 30 kg/m2
  * Patients with a morning serum total testosterone level < 300 ng/dL on at least two separate occasions during the Screening and/or Baseline periods.
  * Patients with inappropriately low gonadotropins at screening given the low testosterone:
* Luteinizing hormone (LH) ≤ ULN
* Follicle stimulating hormone (FSH) ≤ ULN
* Estradiol within or above the normal range (defined as ≥ LLN of the approved assay)

  * Normal hypothalamic/pituitary function, including:
* Prolactin: within the normal range
* Thyroid stimulating hormone (TSH): within the normal range
* Ferritin: within the normal range
* Patients agree to use a barrier method of contraception (e.g., condom), for the duration of the study and for at least 3 months following their Study Completion visit to prevent BGS649 exposure to their partners.

Exclusion Criteria:

* Patients with hypogonadism, not related to obesity or as a result of other underlying issues
* Patients with significant major organ class illness (e.g. kidney or liver disease).
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-08; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Parkin, PhD FRCP, Study Director — Mereo BioPharma
Locations (5):
- United States (4):
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Miramar, Florida
  - Novartis Investigative Site, West Valley City, Utah
- Novartis Investigative Site, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 participants enrolled in Part 1 and 15 participants enrolled in part 2.
Groups:
- BGS649 Part 1: BGS649 1mg and 0.1mg in hard gelatin capsules. In part 1 there was individualised dosing to titrate the subject's testosterone into the normal range. If the dose was lower than 0.1mg then specific instructions for dilution of an oral solution of BGS649 were provided.
- BGS649 Part 2: BGS649 0.3mg hard gelatin capsule given orally on Day 1 and 0.1mg BGS649 capsule on other treatment visits (week 1 to 11).
- Placebo to BGS649: Matching placebo to BGS649 (0.3 and 0.1mg). 0.3mg placebo capsule given on Day 1 and 0.1mg placebo capsule on other treatment visits (week 1 to 11).
Period: Part 1
Arm/Group | BGS649 Part 1 | BGS649 Part 2 | Placebo to BGS649
Started (Part 1) | 14 | 0 | 0
Completed | 13 | 0 | 0
Not Completed | 1 | 0 | 0
Period: Part 2
Arm/Group | BGS649 Part 1 | BGS649 Part 2 | Placebo to BGS649
Started | 0 | 7 | 8
Completed | 0 | 6 | 8
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- BGS649 (Part 2): BGS649 0.3mg hard gelatin capsule given orally on Day 1 and 0.1mg BGS649 capsule on other treatment visits (week 1 to 11).
- Total: Total of all reporting groups
Arm/Group | BGS649 (Part 1) | BGS649 (Part 2) | Placebo to BGS649 (Part 2) | Total
Number analyzed (Participants) | 14 | 7 | 8 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] — Age calculate from date of birth at time of consent Population: Part 1 and Part 2 results were analysed completed separately throughout the study
  years
    Age (Part 1): number analyzed (Participants) | 14 | 0 | 0 | 14
    Age (Part 1) | 50 (9.54) |  |  | 50 (10.1)
    Age (Part 2): number analyzed (Participants) | 0 | 7 | 8 | 15
    Age (Part 2) |  | 51 (10.1) | 50 (11.1) | 50 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Part 1 and Part 2 patients were analysed completed separately throughout the study
  Participants
    Sex (Part 1): number analyzed (Participants) | 14 | 0 | 0 | 14
    Sex (Part 1): Female | 0 |  |  | 0
    Sex (Part 1): Male | 14 |  |  | 14
    Sex (Part 2): number analyzed (Participants) | 0 | 7 | 8 | 15
    Sex (Part 2): Female |  | 0 | 0 | 0
    Sex (Part 2): Male |  | 7 | 8 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Part 1 and Part 2 of the study were reported/analysed separately and so combined totals are not available
  Participants
    Part 1: number analyzed (Participants) | 14 | 0 | 0 | 14
    Part 1: Caucasian | 12 |  |  | 12
    Part 1: Black | 2 |  |  | 2
    Part 1: Native American | 0 |  |  | 0
    Part 2: number analyzed (Participants) | 0 | 7 | 8 | 15
    Part 2: Caucasian |  | 6 | 7 | 13
    Part 2: Black |  | 0 | 1 | 1
    Part 2: Native American |  | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 7 | 8 | 29
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] — Body Mass index calculated Population: Part A and Part B were analysed and reported separately in the study
  kg/m2
    BMI (Part 1): number analyzed (Participants) | 14 | 0 | 0 | 14
    BMI (Part 1) | 34 (3.21) |  |  | 36.6 (4.10)
    BMI (Part 2): number analyzed (Participants) | 0 | 7 | 8 | 15
    BMI (Part 2) |  | 37 (2.9) | 39 (6.2) | 38 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Normal Testosterone Levels
Description: Percentage of patients achieving normal testosterone (2.50 - 9.50 ng/mL) levels at Week 4 and Week 12
Time Frame: At Week 4 and 12
Population: Number/percentage of patients achieving normal sex hormone levels at Week 4 and Week 12 (Part 1 Only)
Measure: Count of Participants; unit: Participants
Arm/Group | BGS649 (Part 1)
Number analyzed (Participants) | 14
Participants
  Week 4 | 14
  Week 12 | 13

2. Primary Outcome: Part 2: Change From Baseline at Homeostatic Model Assessment of Insulin Resistance (HOMA-IR & QUICKI Scores) at Week 4 and 12
Description: Pharmacodynamic change from baseline in HOMA-IR. Score at week 4 and week 12 as an assessment of insulin resistance. Low score representing high insulin sensitivity and a high score representing low insulin sensitivity or insulin resistance. HOMA-IR is a ration of Fasting insulin (mIU/L) : Fasting glucose (mmol). Pharmacodynamic change in QUICKI score at week 4 and week 12 as an assessment of insulin resistance. The QUICKI scale is a log score and a high score representing high insulin sensitivity and low score indicating low insulin sensitivity. Patients with a score below 0.3 are considered diabetic. Week 12 data is missing because there were inaccuracies in dosing of patients and so the study was terminated, only safety data was collected.
Time Frame: Baseline, Week 4 and Week 12
Population: Could not be analysed due to drug administration errors. Week 12 data is missing because they were inaccuracies in the dosing of patients and so the study was terminated early and efficacy data not reported for the affected patients.
Measure: Geometric Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | BGS649 Part 2 | Placebo to BGS649
Number analyzed (Participants) | 7 | 5
units on a scale
  HOMA-IR at 4 weeks | 7.94 [3.72 to 16.92] | 7.45 [2.74 to 20.29]
  QUICKI at 4 weeks | 0.12 [0.11 to 0.14] | 0.13 [0.11 to 0.14]
  HOMA-IR at 12 weeks: number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Part 2: Area Under the Concentration-time Curve From Time Zero to Time 't' (AUC0-168)
Description: PK sampling was performed at 0hr (pre-dose), 1 hr, 8 hr, 24 hr, 72 hr, and 168 hr on the following occasions Week 1, Week 4 and week 11. The AUC 0-168 measures the amount of drug within the subjects blood over the 168h post-dosing at these timepoints.
Time Frame: 11 weeks
Population: PK Analysis Set included 7 patients given BGS649 in Part 2.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | BGS649 (Part 2)
Number analyzed (Participants) | 7
ng*hr/mL
  Week 1 | 114 (36.9)
  Week 4: number analyzed (Participants) | 6
  Week 4 | 152 (48.8)
  Week 11: number analyzed (Participants) | 5
  Week 11 | 167 (21.5)

4. Secondary Outcome: Part 2: Pharmacokinetics of BGS649: Maximum (Peak) Observed Blood Drug Concentration After Single Dose Administration (Cmax)
Description: PK sampling was performed at 0hr (pre-dose), 1 hr, 8 hr, 24 hr, 72 hr, and 168 hr on the following occasions Week 1, Week 4 and week 11.
Time Frame: Week 1 to Week 11
Population: PK Analysis Set
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BGS649 (Part 2)
Number analyzed (Participants) | 7
ng/mL
  Week 1 | 2.83 (0.998)
  Week 4: number analyzed (Participants) | 6
  Week 4 | 1.69 (0.610)
  Week 11: number analyzed (Participants) | 5
  Week 11 | 1.69 (0.261)

5. Secondary Outcome: Part 2: Pharmacokinetics of BGS649: Time to Reach Maximum (Peak) Blood Drug Concentration After Single Dose Administration (Tmax)
Description: as for outcome 4
Time Frame: Week 1 to Week 11
Population: PK Population
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BGS649 (Part 2)
Number analyzed (Participants) | 7
hours
  Week 1 | 1.02 (0.00339)
  Week 4: number analyzed (Participants) | 6
  Week 4 | 1.01 (0.0136)
  Week 11: number analyzed (Participants) | 5
  Week 11 | 0.993 (0.0450)

6. Secondary Outcome: PK of BGS649 Elimination Half-life Associated With the Terminal Slope of a Semi Logarithmic Concentration-time Curve (T1/2)
Description: as for outcome 4
Time Frame: Week 1 to Week 11
Population: PK Analysis Set. Sparse PK sampling (4 samples over 672 h) was included for the PK profile for Week 4; Cmax was included in λz estimation, therefore T1/2 was not reported for all profiles in Week 4.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | BGS649 (Part 2)
Number analyzed (Participants) | 7
hours
  Week 1: number analyzed (Participants) | 6
  Week 1 | 474 (114)
  Week 4: number analyzed (Participants) | 0
  Week 11 | 489 (83)

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Does not differ to clinicaltrials.gov. definitions
Groups:
- BGS649 (Part 1) Open Label: Individualised doses to titrate testosterone levels to within normal range. Doses ranged between 0.003mg and 5mg in total over the 11 week treatment period. For doses below 0.1mg, separate pharmacy instructions were provided to dilute an oral solution of BGS649.
- BGS649 (Part 2): All subjects were given 0.3mg on Day 1 and then 0.1mg on all other dosing visits (weeks 2-11).
- Placebo to BGS649 (Part 2): Matching placebo capsules on Day 1 and all other dosing visits (weeks 2-11).
Arm/Group | BGS649 (Part 1) Open Label | BGS649 (Part 2) | Placebo to BGS649 (Part 2)
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/7 | 1/8
Other Adverse Events (participants affected / at risk) | 11/14 | 5/7 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGS649 (Part 1) Open Label (N=14) | BGS649 (Part 2) (N=7) | Placebo to BGS649 (Part 2) (N=8)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGS649 (Part 1) Open Label (N=14) | BGS649 (Part 2) (N=7) | Placebo to BGS649 (Part 2) (N=8)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Spontaneous penile erection (Reproductive system and breast disorders) | 4 (4) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1 (1)
Oropharyngeal pain (Reproductive system and breast disorders) | 3 (3) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Asthenia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Increased appetitie (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
Libido increased (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Stress (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Terminal insomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Part 2 of the study was early terminated due to incorrect dosing, therefore only 8 of the 15 subjects enrolled completed 11 doses of treatment, and the remaining 7 subjects had incomplete dosing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs must seek written permission from the sponsor prior to publication of any trial results.